CLINICAL TRIAL: NCT04817917
Title: Seroprevalence of Neutralizing Antibodies Against Japanese Encephalitis Virus Among 6 Years Old Children With 5 Different Immunization Strategies in Zhejiang Province, China: An Open-labeled, Ambidirectional Cohort Study
Brief Title: Seroprevalence of Neutralizing Antibodies Against Japanese Encephalitis Virus Among 6 Years Old Children With 5 Different Immunization Strategies in Zhejiang Province
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Collaborators: Liaoning Chengda Biotechnology CO., LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZJCDC20210317
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-07

CONDITIONS: Japanese Encephalitis; Vaccine Preventable Disease; Vaccine Reaction
Keywords: Japanese Encephalitis; Seroprevalence; Immunogenicity; Immunization schedule; Safety
MeSH Terms: conditions — Encephalitis, Japanese; Vaccine-Preventable Diseases | interventions — Japanese Encephalitis Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 3JEV-I (Group 1) (Experimental): Retrospective: 3 doses of JE vaccines. 2 doses of Inactivated JE Vaccine (JEV-I, 7-10 days apart) at 8 months of age and 1 dose of JEV-I at 2 years old.
  Prospective: 1 booster dose of JEV-I at 6 years old.
  Interventions: Biological: Japanese Encephalitis Vaccine (Vero Cell), Inactivated;
- JEV-L+JEV-I (Group 2) (Experimental): Retrospective: 2 doses of JE vaccines.
  1 dose of JE attenuated live vaccine (JEV-L) at 8 months of age and 1 dose of JEV-I at 2 years old.
  Prospective: 1 booster dose of JEV-I at 6 years old.
  Interventions: Biological: Japanese Encephalitis Vaccine (Vero Cell), Inactivated;
- JEV-L+2JEV-I (Group 3) (Experimental): Retrospective: 3 doses of JE vaccines.
  1 dose of JEV-L at 8 months of age and 2 dose (7-10 days apart) of JEV-I at 2 years old.
  Interventions: Other: No prospective interventions
- 2JEV-I+JEV-L (Group 4) (Experimental): Retrospective: 3 doses of JE vaccines. 2 doses of JEV-I (7-10 days apart) at 8 months of age and 1 dose of JEV-L at 2 years old.
  Interventions: Other: No prospective interventions
- 2JEV-L (Group 5) (Experimental): Retrospective: 2 doses of JE vaccines. 2 doses of JEV-L respectively administered at 8 months of age and 2 years old.
  Interventions: Other: No prospective interventions

INTERVENTIONS:
Biological: Japanese Encephalitis Vaccine (Vero Cell), Inactivated; — The investigators recruit 6 years old children who have been vaccinated by 2-3 doses of JE vaccines with different immunization strategies. For participants from Group 1 and Group 2 who haven't completed the JE immunization schedules, a booster dose of JEV-I will be administered at 6 years old.
  Arms: 3JEV-I (Group 1); JEV-L+JEV-I (Group 2)
Other: No prospective interventions — The investigators recruit 6 years old children who have been vaccinated by 2-3 doses of JE vaccines with different immunization strategies. Participants from Group 3-5 have completed the JE immunization schedules with JEV-I or/and JEV-L. No prospective intervention will be given.
  Arms: 2JEV-I+JEV-L (Group 4); 2JEV-L (Group 5); JEV-L+2JEV-I (Group 3)

SUMMARY:
This study is to evaluate the seroprevalence of neutralizing antibodies against Japanese encephalitis (JE) virus in children aged 6 years who were previously administered with 5 different immunization strategies by JE attenuated live vaccine (JEV-L) or/and inactivated vaccine (JEV-I). The secondary objective is to evaluate the immunogenicity of the booster dose of JEV-I at 6 years old for those previously immunized with 3 doses of JEV-I or those sequential administered with 1 dose of JEV-L and another dose of JEV-I.

DETAILED DESCRIPTION:
Based on the retrospective registry in Zhejiang Provincial Immunization Information System, healthy children aged 6 years from 5 cohorts were included according to their previous immunization schedules on JE: 3 doses of JEV-I (Group 1), JEV-L+ JEV-I (Group 2), JEV-L+ JEV-I + JEV-I (Group 3), JEV-I + JEV-I+ JEV-L (Group 4), and 2 doses of JEV-L (Group 5). According to immunization programs in China, a booster dose of JEV-I is needed at the age of 6 for Group 1 and Group 2. A pre-vaccination blood sample (2.5ml) will be collected to evaluate the proportions of seropositivity before the booster dose of JEV-I. A second blood sample will be collected 28-35 days after the booster dose. Immunogenicity of the booster dose will be assessed by seroconversion rates, proportions of seropositivity and GMTs for these two groups. In addition, safety will be assessed with the occurrence of adverse events reported in these two groups. For the rest three groups who have completed the immunization schedules on JE, only one blood sample will be taken at the age of 6 to evaluate the proportions of seropositivity and GMTs after 4 years post the complete immunization schedules. Plague reduction neutralization test (PRNT) against both vaccine strains (SA-14-14-2 strain for JEV-L and Beijing P3 strain for JEV-I) will be used to test neutralizing antibody titers, so as to avoid potential bias in favor of either vaccine. PRNT50 titers (the reciprocal of the serum dilution that reduced the virus plaque count by 50% compared with the virus-only controls) ≥ 1:10 are deemed as positive.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥ 72 months to < 75 months.
* Participants have completed routine immunization schedules in time.
* Participants are healthy native residents.
* Parents/guardians can understand the protocol requirements, provide informed consent, accept all scheduled visits, and comply with all trial procedures.

Exclusion Criteria:

* History of neurological diseases or related symptoms.
* An acute illness with fever (temperature ≥ 37.1℃) or any acute onset of chronic diseases.
* Known impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin in the past 3 months.
* Known allergy to any constituent of the vaccine.
* Have been injected with other vaccines or any clinical trial drugs in the past 4 weeks.
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the vaccine.

Ages: 72 Months to 75 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 712 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportions of seropositivity of neutralizing antibodies against JE at the age of 6 | At the age of 6. Test immediately after enrollment by a dose of blood sample.
  Defined as any positive antibody (neutralizing antibody titers ≥1:10) response in children aged 6.
Geometric Mean Titers (GMTs) or Median antibody titers for children aged 6 years | At the age of 6. Test immediately after enrollment by a dose of blood sample.
  Neutralizing antibody titers by plaque-reduction neutralization tests (PRNT).

SECONDARY OUTCOMES:
Seroconversion rates of the booster dose of JEV-I for Group 1 and Group 2 | before and 28-35 days after the booster dose.
  Defined as any positive antibody (neutralizing antibody titers ≥1:10) response in children who were seronegative prior to the booster dose, or at least a four-fold increase for children who had pre-existing positive antibodies.
Proportion of seropositivity of neutralizing antibodies against JE after the booster dose for Group 1 and Group 2. | 28-35 days after the booster dose.
  Defined as any positive antibody (neutralizing antibody titers ≥1:10) response after the booster dose.
Geometric Mean Titers (GMTs) or Median antibody titers after the booster dose for Group 1 and Group 2. | 28-35 days after the booster dose.
  Neutralizing antibody titers by PRNT.
Safety of the booster dose for Group 1 and Group 2 | From inoculation to 30 days after the inoculation.
  The occurrence of adverse events for the booster dose

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Liandu center for disease control and prevention, Lishui, Zhejiang
  - Kecheng center for disease control and prevention, Quzhou, Zhejiang
  - Pingyang center for disease control and prevention, Wenzhou, Zhejiang